CLINICAL TRIAL: NCT02037386
Title: H-Side Branch Stent, A New Stent for the Treatment of True Bifurcation Lesions
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: problem with balloon catheter
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2011-0096
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Coronary Artery Disease
Keywords: Side branch stent; Coronary bifurcation lesion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- H-side branch stent (Experimental): H-side branch stent group
  Interventions: Device: H-side branch stent

INTERVENTIONS:
Device: H-side branch stent — Implantation of H-side branch stent at coronary bifurcation stenotic lesion

SUMMARY:
Intervention for coronary bifurcation lesion is about 10~20% of entire percutaneous coronary intervention (PCI). Bifurcation lesion is difficult to be treated and prognosis of PCI at bifurcation lesion has been poorer compared to that at non-bifurcation lesion. Furthermore, occlusion of side branch frequently occurred during PCI. Several techniques to prevent occlusion of side branch have been developed, but outcomes are not to be satisfied. H-side branch stent is developed to treat coronary side branch lesion and composed of proximal, connecting and distal parts. In vivo study performed in pigs showed effective H-side branch stent. This study is to confirm safety and efficacy of H-side branch stent for treatment of coronary side branch lesion.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years old
* Patient with angina or asymptomatic ischemic cardiomyopathy who is required to be treated with stent at coronary bifurcation lesion
* Bifurcation lesion with 2.5~4.0mm of main vessel diameter, <30mm of main vessel length and ≥2.0mm of branched vessel diameter

Exclusion Criteria:

* Acute myocardial infarction
* Confirmed or suspicious presence of thrombus in target lesion
* In-stent restenosis lesion
* Visual angulation with ≥75°
* Lesion with severe calcification or severe tortuosity
* Left main lesion
* Chronic total occlusion lesion
* Graft lesion
* Contraindication to antiplatelet drugs
* Left ventricular dysfunction (LVEF ≤40%)
* Severe hepatic dysfunction (≥2.5 times than reference of AST or ALT)
* Renal dysfunction (serum Creatinine > 2.0mg/dL)
* History of cerebral hemorrhage, pulmonary or gastrointestinal bleeding
* Hypersensitivity of aspirin, clopidogrel or contrast media
* Pregnant woman or possibility of pregnancy during clinical study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | During 6 months after implantation of H-side branch stent
  composite of cardiovascular death, non-fatal myocardial infarction, stent thrombosis, target lesion revascularization

REFERENCES:
- [Background] Hong MK, Shim JM, Youn YJ, Lee KH, Kim JS, Ko YG, Lee SH, Choi D, Yoon J, Jang Y. A new stent design for the treatment of true bifurcation lesions: H-side branch stents. J Interv Cardiol. 2010 Feb;23(1):54-9. doi: 10.1111/j.1540-8183.2009.00519.x. Epub 2009 Dec 17. PMID 20040003